CLINICAL TRIAL: NCT00560326
Title: A Long-term, Non-comparative Study to Evaluate the Safety and Efficacy of Tacrolimus Oint¬Ment in Paediatric Patients
Brief Title: Tacrolimus Ointment Long Term Safety in Young Children With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-06-33
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: Paediatric patients; Tacrolimus; Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Tacrolimus Ointment 0.03%

INTERVENTIONS:
Drug: Tacrolimus Ointment 0.03% — Once or twice daily topical application
  Other Names: Protopic 0.03%

SUMMARY:
The objective of this study is to assess the safety and efficacy of 0.03% tacrolimus ointment as long-term treatment in paediatric patients with atopic dermatitis.

DETAILED DESCRIPTION:
This is a long-term, multi-centre, non-comparative phase II study. All centres participating in the FG-506-06-32 pharmacokinetics study will be offered the protocol as a follow-up. Only patients enrolled by those centres for the above mentioned study, who applied at least one dose of study medication and benefited from treatment with 0.03% tacrolimus ointment, can be enrolled.

During episodes of active disease, a thin coat of ointment is applied on each lesion. In the first three weeks, frequency of application is twice a day; after three weeks treatment is continued once a day. All atopic dermatitis lesions are treated until clearance (i.e. itch has gone). In case of a flare-up or worsening treatment twice daily treatment is re-started for three weeks and thereafter reduced to once daily.

Safety is assessed from adverse events reported by the patient and/or his parents or observed by the investigator at the site of application and elsewhere. The safety evaluation includes monitoring of routine haematology and serum chemistry parameters. Blood samples are analysed by local laboratories. Blood samples are taken to determine concentrations of tacrolimus.

Height, weight and pulse of the patient are recorded at each visit.

Efficacy is assessed by physician's global evaluation of clinical response, patient's parent/guardian's assessment of global response, physician's assessment of individual signs and the affected area assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has participated in the study FG-506-06-32, has applied at least one dose of study medication and has benefited from treatment in the opinion of the investigator.
* Patient is likely to benefit from further treatment with tacrolimus ointment in the opinion of the investigator.

Exclusion Criteria:

* Patient has a skin disorder on the affected (and to be treated) area, other than atopic dermatitis, requiring treatment.
* Patient has clinically infected atopic dermatitis.

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2003-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Assess safety from observations of adverse events, laboratory examinations, pulse, height, weight and tacrolimus blood concentrations | 24 months

SECONDARY OUTCOMES:
Assess efficacy from parameters as follows: - Physician's global evaluation of clinical response - Physician's assessment of individual signs - Affected area - Parent/guardian's assessment of global response - EASI | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (8):
- Canada (3):
  - Halifax
  - Vancouver
  - Waterloo
- Helsinki, Finland
- Ireland (2):
  - Drogheda
  - Dublin
- Riga, Latvia
- London, United Kingdom